CLINICAL TRIAL: NCT02756728
Title: A Randomized Phase I/II Study of BI-505 in Conjunction With High-dose Melphalan and Autologous Stem Cell Transplantation for Multiple Myeloma
Brief Title: A Phase I/II Study of BI-505 in Conjunction With Autologous Stem Cell Transplant in Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Full clinical hold from FDA
Sponsor: BioInvent International AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-BI-505-03
Record Dates: First submitted 2016-04-18; First posted 2016-04-29 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HDM+ASCT (Active Comparator): Standard of care; High dose Melphalan + Autologous Stem Cell Transplantation
  Interventions: Other: High dose melphalan; Other: Autologous stem cell transplantation
- BI-505 (Experimental): Biweekly infusions of BI-505 in addition to High dose Melphalan + Autologous Stem Cell Transplantation
  Interventions: Biological: BI-505; Other: High dose melphalan; Other: Autologous stem cell transplantation

INTERVENTIONS:
Biological: BI-505 — Treatment with BI-505 10 mg/kg bi-weekly infusion, up to 9 doses over 4 months
  Arms: BI-505
Other: High dose melphalan — High dose melphalan (HDM)
Other: Autologous stem cell transplantation — Autologous stem cell transplantation (ASCT)

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of administering BI-505 in conjunction with high dose melphalan and stem cell transplantation in multiple myeloma patients.

DETAILED DESCRIPTION:
N/A study is closed

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of multiple myeloma by 2014 IMWG criteria and have been recommended to undergo HDM + ASCT as a standard-of-care therapy for their multiple myeloma.
* Subjects must have adequate vital organ function and functional status for HDM + ASCT
* Subjects must have collected and cryopreserved ≥4x106 hematopoietic stem cells per kg of actual body weight that are suitable for use in autologous stem cell transplantation in the judgment of the investigator.
* At the time of enrollment, subjects must have had at least a partial response, as defined by IMWG criteria and in comparison to baseline/pre-treatment parameters, to an induction regimen containing lenalidomide and/or bortezomib.
* Subjects must have measurable disease according to one of the following criteria:

  1. Serum M-spike ≥0.1 g/dl
  2. Urine M-spike >200 mg in a 24-hour urine collection
  3. Involved serum free light chain above the upper limit of normal and a serum free light chain ratio outside the normal range.
* At the time of enrollment, subjects must be within 12 months of the first dose of initial/induction therapy, and the anticipated day of ASCT must be within 12 months of the first dose of initial/induction therapy

Exclusion Criteria:

* Prior allogeneic or autologous hematopoietic stem cell transplant
* Current active infections, including HIV and hepatitis C and B
* Autoimmune disease requiring ongoing immunosuppressive therapy.
* History of atrial fibrillation or flutter, including paroxysmal atrial fibrillation or flutter.
* History of transient ischemic attack or stroke.
* At the time of enrollment, subjects must not have required multi-agent continuous-infusion cytotoxic chemotherapy (e.g., regimens such as D-PACE) as part of their initial/induction therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Determine the safety and feasibility of administering BI-505 in conjunction with HDM+ASCT in multiple myeloma patients | Adverse events will be assessed within 30 days of ASCT in the safety part of the study.
  UNK
Phase II: Determine the effect of BI-505 on rate of stringent complete response for multiple myeloma patients with measurable disease pre-ASCT. | At Day 100 after ASCT
  UNK

SECONDARY OUTCOMES:
Determine the effect of BI-505 on rate of stringent complete response (sCR) at day 100 in subgroups stratified according to response to initial therapy (+/- VGPR). | Day 100 after ASCT
  UNK
Determine the effect of BI-505 administered in conjunction with HDM + ASCT on IMWG response category (PR, VGPR, CR, sCR) at one year post-ASCT and progression-free survival. | At one year and up to three years after ASCT
  UNK
Evaluate the effect of BI-505 on MRD-negative rate at day 100 and change in MRD status at day 100 compared to baseline. | Day 100
  UNK
Evaluate anti-myeloma effect of BI-505 monotherapy, prior to HDM + ASCT | Prior to HDM + ASCT (from Day -17 until Day 0)
  UNK
Evaluate bone marrow immune cell composition and phenotype, including macrophage infiltration and expression of intracellular adhesion molecule (ICAM)-1 expression on multiple myeloma plasma cells, as potential biomarkers of response to BI-505 | Day 100 compared to Baseline (Day -17 and Day -2)
  UNK
Evaluate the pharmacokinetic profile of BI-505 in this clinical setting by analysing Cmax | All dosing visits throughout the study (up to 9 biweekly infusions of BI-505). Day -17, day -3, day 11, day 25, day 39, day 53, day 67, day 81, day 95, day 123
  Maximum Plasma Concentration (Cmax)
Evaluate the pharmacokinetic profile of BI-505 in this clinical setting by analysing Tmax | All dosing visits throughout the study (up to 9 biweekly infusions of BI-505). Day -17, day -3, day 11, day 25, day 39, day 53, day 67, day 81, day 95, day 123
  Time to reach Cmax (Tmax)
Evaluate the pharmacokinetic profile of BI-505 in this clinical setting by analysing AUC | All dosing visits throughout the study (up to 9 biweekly infusions of BI-505). Day -17, day -3, day 11, day 25, day 39, day 53, day 67, day 81, day 95, day 123
  Area under the curve (AUC)
Evaluate the pharmacokinetic profile of BI-505 in this clinical setting by analysing CL | All dosing visits throughout the study (up to 9 biweekly infusions of BI-505). Day -17, day -3, day 11, day 25, day 39, day 53, day 67, day 81, day 95, day 123
  Clearance (CL)
Evaluate the pharmacokinetic profile of BI-505 in this clinical setting by analysing Vss | All dosing visits throughout the study (up to 9 biweekly infusions of BI-505). Day -17, day -3, day 11, day 25, day 39, day 53, day 67, day 81, day 95, day 123
  Volume of distribution at steady state (Vss)
Evaluate the pharmacokinetic profile of BI-505 in this clinical setting by analysing t1/2 | All dosing visits throughout the study (up to 9 biweekly infusions of BI-505). Day -17, day -3, day 11, day 25, day 39, day 53, day 67, day 81, day 95, day 123
  Elimination half-life (t1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Garfall, MD, Principal Investigator — Div of Hema/Onc, Dept.of Med, Perelman Center Advanced Med, Philadelphia PA
Locations (1):
- Perelman School of Medicine/Hospital of the Univ. of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No